CLINICAL TRIAL: NCT04716881
Title: A Bioequivalence Study Comparing Vivitrol and O'Neil Long Acting Naltrexone Implant (OLANI) in Healthy Participants
Brief Title: Pharmacokinetic Study of Vivitrol in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Go Medical Industries Pty Ltd (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); New York State Psychiatric Institute (Other); Columbia University (Other); Clinilabs, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GM0019; UG3DA047720 (NIH); 406190 (Other: NIH ERA Human Subjects Study Number)
Record Dates: First submitted 2021-01-17; First posted 2021-01-20 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Opioid-use Disorder
Keywords: naltrexone; opioids; Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vivitrol (naltrexone) (Experimental): Intramuscular injection of Vivitrol (naltrexone), 380 mg. Six doses given 28 days apart.
  Interventions: Drug: Naltrexone 380 MG

INTERVENTIONS:
Drug: Naltrexone 380 MG — Vivitrol (naltrexone) 380 mg delivered intramuscularly every 28 days
  Other Names: Vivitrol

SUMMARY:
This is a Phase I, single-center, single arm, open-label study, to establish the pharmacokinetic (PK) parameters of Vivitrol 380 mg IM injection (IP), a US Food and Drug Administration (FDA) approved medication.

DETAILED DESCRIPTION:
This is a Phase I, single-center, single arm, open-label study, to establish the PK parameters of Vivitrol 380 mg IM injection (IP), a US FDA approved medication. Participants will be healthy volunteers with no significant medical or mental health disorders, who have completed participation in clinical trial GM0017 (i.e. have received the OLANI treatment and have subsequently provided two consecutive plasma levels of naltrexone (NTX) <0.1ng/mL).

This study will examine the PK profile of Vivitrol IM 380 mg over 6 doses for a treatment period of 196 days. Intense sampling will occur after the 1st and 6th dose of Vivitrol. Participants will be without a DSM 5 - Substance Related Disorders classification. Participants will be required to undergo a Naloxone Challenge Test (NCT) to confirm opiate naivety before administration of the IP. No randomization will occur.

ELIGIBILITY:
Inclusion Criteria:

* Have completed GM0017 (i.e. been administered OLANI (3.6 gram) and provided two consecutive monthly blood samples of NTX below 0.1 ng/mL)
* Men or women between ≥18 and <58 years old Without DSM 5 - Substance Related Disorders classification; in sustained remission is not exclusionary
* Able and willing to comply with the requirements of the protocol
* Able and willing to provide written informed consent
* Willing to undergo an injection of NTX to allow for investigational drug administration in the intramuscular tissue
* Have an initial weight between 45.3 and 81.6 kilograms (inclusive) or have a BMI inclusive of 18.5 to 30.0.

Exclusion Criteria:

* Is currently on active NTX medication.
* Positive UDS at screening for illicit substances.
* Has a condition which requires treatment with opioid based medication.
* Has a known hypersensitivity to NTX.
* Is prone to skin rashes, irritation or has a skin condition such as recurrent eczema that is likely to impact the injection site area, or as determined by the evaluating physician.
* Demonstrates any abnormal skin tissue in the proposed injection area.
* Is pregnant or planning to be. Women need to have negative pregnancy test at screening. Women need to agree to practice an effective method of contraception throughout participation.
* Participant is breastfeeding or planning to be.
* Has a current significant neurological (including cognitive and psychiatric disorders),
* Any clinically important abnormal finding as determined by medical history, physical examination, ECG or clinical laboratory tests.
* Any additional condition(s) that in the investigator's opinion would prohibit the participant from completing the study or would not be in the best interest of the participant.
* ALT or AST >3 times the upper end of the laboratory normal range.
* Any methadone use 14 days prior to screening, and up to Study Day 0.
* Current DSM 5 diagnosis of schizophrenia, bipolar, anxiety, or depressive disorder, confirmed by MINI assessment, or currently treated with medications for anxiety or depression. Past history (in remission DSM 5 classification) of anxiety or depression is not exclusionary.
* Any elevated risk for suicide measured using the Columbia Suicide Severity Rating Scale, endorsing any of the items in the past month (C-SSRS, Lifetime)
* Is participating or intending to participate in any other clinical trial during the duration of this study.
* Is allergic to any of the ingredients in Vivitrol or the diluent used to mix Vivitrol (i.e. carboxymethylcellulose sodium, polysorbate 20, sodium chloride, sodium hydroxide and hydrochloric acid as pH adjusters, in water for injection).

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vivitrol (Naltrexone)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50.0 [40 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9
Body Mass Index (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 25.90 [22.8 to 29.9]

OUTCOME MEASURES:

1. Primary Outcome: Median Cmax of Naltrexone (After 1st Dose)
Description: Single-dose PK measurement of the maximum observed plasma naltrexone concentration (Cmax) after dosing on Day 0
Time Frame: 1st dose: Day 0 (predose), 1, 2, 4, 8, 12 hours, 24 hours (Day 1), Days 1.5, 1.75, 2, 3, 5, 7, 10, 14, 17, 21, 24, and 28.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 14.10 [13.40 to 23.10]

2. Primary Outcome: Median Tmax of Naltrexone (After 1st Dose)
Description: Single-dose PK measurement of the time to maximum plasma naltrexone concentration (Tmax) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day | 2.00 [1.96 to 3.02]

3. Primary Outcome: Median AUC0-inf of Naltrexone (After 1st Dose)
Description: Single-dose PK measurement of the area under the plasma concentration-time curve for naltrexone from time 0 extrapolated to infinity (AUC0-inf) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day*ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day*ng/mL | 153.00 [107.01 to 180.83]

4. Primary Outcome: Median Ctrough of Naltrexone (After 1st Dose)
Description: Single-dose PK measurement of naltrexone concentration at the end of the dosing interval (Ctrough) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 0.81 [0.49 to 1.06]

5. Primary Outcome: Median Cmax of 6β-naltrexol (After First Dose)
Description: Single-dose PK measurement of the maximum observed plasma 6β-naltrexol concentration (Cmax) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 20.50 [17.30 to 26.10]

6. Primary Outcome: Median Tmax of 6β-naltrexol (After 1st Dose)
Description: Single-dose PK measurement of the time to maximum plasma 6β-naltrexol concentration (Tmax) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day | 3.02 [2.00 to 3.15]

7. Primary Outcome: Median AUC0-inf of 6β-naltrexol (After 1st Dose)
Description: Single-dose PK measurement of the area under the plasma concentration-time curve for 6β-naltrexol from time 0 extrapolated to infinity (AUC0-inf) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day*ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day*ng/mL | 270.16 [216.32 to 342.38]

8. Primary Outcome: Median Ctrough of 6β-naltrexol (After 1st Dose)
Description: Single-dose PK measurement of 6β-naltrexol concentration at the end of the dosing interval (Ctrough) after dosing on Day 0
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 1.71 [1.33 to 1.97]

9. Primary Outcome: Median Cmax of Naltrexone (After 6th Dose)
Description: PK measurement of the maximum observed plasma naltrexone concentration (Cmax) after 6th dose on Day 140
Time Frame: 6th dose: Day 140 (1, 2, 4, 8 & 12 hours), 141, 141.5, 141.75, 142, 143, 145, 147, 150, 154, 157, 161, 164, 168, 182 and 196
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 14.00 [11.80 to 17.60]

10. Primary Outcome: Median Tmax of Naltrexone (After 6th Dose)
Description: PK measurement of the time to maximum plasma naltrexone concentration (Tmax) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day | 2.00 [1.97 to 2.94]

11. Primary Outcome: Median AUC0-inf of Naltrexone (After 6th Dose)
Description: PK measurement of the area under the plasma concentration-time curve for naltrexone from time 0 extrapolated to infinity (AUC0-inf) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: day*ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day*ng/mL | 167.14 [127.03 to 199.65]

12. Primary Outcome: Median Ctrough of Naltrexone (After 6th Dose)
Description: PK measurement of naltrexone concentration at the end of the dosing interval (Ctrough) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 1.37 [0.52 to 1.75]

13. Primary Outcome: Median Cmax of 6β-naltrexol (After 6th Dose)
Description: PK measurement of the maximum observed plasma 6β-naltrexol concentration (Cmax) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 24.70 [19.50 to 31.00]

14. Primary Outcome: Median Tmax of 6β-naltrexol (After th Dose)
Description: PK measurement of the time to maximum plasma 6β-naltrexol concentration (Tmax) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day | 2.95 [2.00 to 3.02]

15. Primary Outcome: Median AUC0-inf of 6β-naltrexol (After 6th Dose)
Description: PK measurement of the area under the plasma concentration-time curve for 6β-naltrexol from time 0 extrapolated to infinity (AUC0-inf) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: day*ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
day*ng/mL | 310.49 [217.12 to 367.51]

16. Primary Outcome: Median Ctrough of 6β-naltrexol (After 6th Dose)
Description: PK measurement of 6β-naltrexol concentration at the end of the dosing interval (Ctrough) after dosing on Day 140
Time Frame: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ng/mL | 2.02 [1.45 to 3.50]

17. Secondary Outcome: Adverse Events (AEs)
Description: Proportion of participants reporting AEs
Time Frame: Up to Day 196
Measure: Count of Participants; unit: Participants
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 8
Participants | 4

18. Secondary Outcome: Naltrexone Accumulation Ratio (AR) for Cmax
Description: The naltrexone AR was determined for Cmax by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 0.96 (49.16)

19. Secondary Outcome: Naltrexone Accumulation Ratio (AR) for Ctrough
Description: The naltrexone AR was determined for Crough by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 1.58 (33.91)

20. Secondary Outcome: Naltrexone Accumulation Ratio (AR) for AUC0-inf
Description: The naltrexone AR was determined for AUC0-inf by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 1.08 (12.27)

21. Secondary Outcome: 6β-naltrexol Accumulation Ratio (AR) for Cmax
Description: The 6β-naltrexol AR was determined for Cmax by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 1.08 (0.63)

22. Secondary Outcome: 6β-naltrexol Accumulation Ratio (AR) for Ctrough
Description: The 6β-naltrexol AR was determined for Ctrough by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 1.37 (34.53)

23. Secondary Outcome: 6β-naltrexol Accumulation Ratio (AR) for AUC0-inf
Description: The 6β-naltrexol AR was determined for AUC0-inf by dividing the PK parameter for Dose 6 by the PK parameter for Dose 1.
Time Frame: 196 days after the 6th dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Vivitrol (Naltrexone)
Number analyzed (Participants) | 7
ratio | 1.14 (7.43)

ADVERSE EVENTS:
Time Frame: 196 days
Arm/Group | Vivitrol (Naltrexone)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivitrol (Naltrexone) (N=8)
Injection site inflammation (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (2)
Corona virus infection (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Aborted pregnancy (Social circumstances) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT04716881/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT04716881/ICF_001.pdf